CLINICAL TRIAL: NCT04236609
Title: ABILITY Diabetes Global
Brief Title: Randomized Comparison of Abluminus DES+ Sirolimus-Eluting Stents Versus Everolimus-Eluting Stents in Coronary Artery Disease Patients With Diabetes Mellitus Global
Acronym: ABILITY
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Concept Medical Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: COMED.CT.DES.001
Record Dates: First submitted 2020-01-15; First posted 2020-01-22 (Actual); Last update posted 2023-03-27 (Actual); Status verified 2023-03

CONDITIONS: Diabetes; Coronary Artery Disease; Acute Coronary Syndrome
MeSH Terms: conditions — Diabetes Mellitus; Coronary Artery Disease; Acute Coronary Syndrome

STUDY DESIGN:
Intervention Model Description: Target lesions should be treated in accordance with the randomization schedule after meeting the clinical and angiographic inclusion and exclusion criteria following the instruction for use of the study stent.
  Additional lesions (other vessels) may be staged up to 45 days post-index procedure but must be treated with the same stent.
  Dual antiplatelet therapy must be prescribed in alignment with the Instructions for Use of the DES and the guidelines
Who Masked: Care Provider, Outcomes Assessor
Masking Description: The staff (i.e. research nurses, research coordinators and other practitioners) involved in the follow-up care of study subjects and the Clinical Events Committee (CEC) adjudicators will be blinded to the patient assignment;
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Abluminus DES+ sirolimus- eluting stents (SES) (Active Comparator): Enrolled patients will undergo angioplasty with Abluminus DES+ sirolimus- eluting stents (SES) and will be followed for two years. The DES procedure will be conducted in accordance with the CE mark instructions for use for the Abluminus DES+ sirolimus- eluting stents (SES).
  Interventions: Device: Abluminus DES+ Sirolimus Eluting Stent System (SES)
- XIENCE Everolimus-Eluting Stents (EES) (Active Comparator): Enrolled patients will undergo angioplasty with XIENCE Everolimus-Eluting Stents (EES) and will be followed for two years. The DES procedure will be conducted in accordance with the CE mark instructions for use for the XIENCE Everolimus-Eluting Stents (EES).
  Interventions: Device: XIENCE Everolimus Eluting Coronary Stent System (XIENCE family)

INTERVENTIONS:
Device: Abluminus DES+ Sirolimus Eluting Stent System (SES) — The Sirolimus-eluting stent manufactured by Envision and distributed by Concept Medical
  Arms: Abluminus DES+ sirolimus- eluting stents (SES)
Device: XIENCE Everolimus Eluting Coronary Stent System (XIENCE family) — The Everolimus-eluting stent manufactured and distributed by Abbott Vascular Santa Clara, CA
  Arms: XIENCE Everolimus-Eluting Stents (EES)

SUMMARY:
To compare in diabetic patients eligible for percutaneous coronary intervention (PCI) with minimal exclusion criteria, the efficacy and safety of Abluminus DES+ sirolimus- eluting stents (SES) versus XIENCE Everolimus-Eluting Stents (EES). At least 40% of patients are expected to be affected by multivessel coronary artery disease and 30% with acute coronary syndrome

DETAILED DESCRIPTION:
This study aims to determine which DES will best treat the diabetic population. Specifically, the research question of this trial is to evaluate the use of a novel sirolimus-eluting stent coated with drug-eluting polymer after crimping on the balloon as compared to the standard-of-care EES in the treatment of de novo coronary artery disease in patients with diabetes mellitus. ABILITY is a prospective, multi-center, multinational, randomized, open label, 2-arm parallel group, post-approval study.

ELIGIBILITY:
Inclusion Criteria:

Clinical Inclusion Criteria

1. Patient understands the trial requirements and the treatment procedures and provides written informed consent;
2. Age ≥ 18 years of age (> 19 years of age for South Korea and ≥ 21 years of age for Singapore);
3. Diabetic patient: either:

   1. Patient with a previous documented diagnosis of diabetes mellitus (Type 1 or Type 2) and currently undergoing pharmacological treatment (oral hypoglycemic agents or insulin)
   2. Newly diagnosed diabetes: either:

   i. Fasting plasma glucose (FPG) ≥126 mg/dL (7.0 mmol/L). Fasting is defined as no caloric intake for ≥8 hours1 or ii. Two-hour plasma glucose ≥200 mg/dL (11.1 mmol/L) following a 75g oral glucose tolerance test or iii. HbA1c level ≥ 7% (53 mmol/mol) Patients who are newly diagnosed are included even if they are not on pharmacological treatment (oral hypoglycemic agents or insulin)
4. Symptomatic coronary artery disease including chronic stable angina, silent ischemia, and non-ST-segment elevation acute coronary syndrome (NSTE-ACS)
5. Patient is eligible for percutaneous coronary intervention (PCI); Previous PCI (with balloon angioplasty or stenting) is allowed if performed >12 months before index procedure;
6. Patient is willing and able to comply with all protocol-required follow-up evaluations.

   Angiographic Inclusion Criteria (visual estimate)
7. Presence of ≥1 de novo coronary artery stenosis >50% in a native coronary artery which can be treated with a stent ranging in diameter from 2.25 to 4.0 mm and can be covered with 1 or multiple stents; and
8. No limitation to the number of treated lesions, number of vessels, or lesion length if the patient is judged eligible for PCI by the treating physician according to the local standard of care.

Exclusion Criteria:

Clinical Exclusion Criteria

1. Patient lacking capacity (i.e. patient suffering from dementia and others) to provide informed consent
2. Patient in cardiogenic shock;
3. Patient has known allergy to the study stent system or protocol-required concomitant medications (e.g. aspirin, clopidogrel, prasugrel, ticagrelor, heparin, stainless steel, platinum, chromium, sirolimus, everolimus, radiographic contrast material) that cannot be adequately pre-medicated;
4. Planned surgery (cardiac and non-cardiac) within 6 months after the index procedure unless the dual-antiplatelet therapy (DAPT) can be maintained throughout the peri-surgical period;
5. Patient undergoing primary percutaneous coronary intervention for ST-segment elevation myocardial infarction (STEMI)
6. Patient is pregnant, nursing, or is a woman of child-bearing potential who is not surgically sterile, < 2 years postmenopausal, or does not consistently use effective methods of contraception*;
7. Patient has any other serious medical illness (e.g., cancer, end-stage congestive heart failure) that may reduce life expectancy to less than 12 months;
8. Acute or chronic renal dysfunction (creatinine >3.0 mg/dl);
9. Currently participating in another investigational drug or device study.

   Angiographic Exclusion Criteria
10. In-stent restenotic lesions;
11. Lesions involving venous or arterial bypass grafts.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3050 (Actual)
Dates: Start 2020-06-15 (Actual); Primary Completion 2023-10-30 (Estimated); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
Rate of Ischemia-driven TLR | 1 year FU
  powered for non-inferiority and sequentially superiority
Rate of Target lesion failure TLF | 1 year FU, powered for non-inferiority
  composite of cardiovascular death, target vessel myocardial infarction [MI], or ischemia driven target lesion revascularization [idTLR])

SECONDARY OUTCOMES:
Safety composite endpoint | 1 year (non-inferiority)
  Safety composite endpoint of the occurrence of cardiovascular death and target-vessel myocardial infarction (MI)
co-primary TLR endpoint | 2 Year FU
  In case the co-primary TLR endpoint (TLR for non-inferiority) will be demonstrated at 1 year, then the occurrence of ischemia-driven TLR at 2-year FU will be evaluated (efficacy endpoint - superiority)
Composite of cardiovascular death, target vessel MI and ischemia-driven TLR (TLF) | 1 year FU
  Cardiovascular death is defined as death resulting from cardiovascular causes. The following categories may be collected:
  1. Death caused by acute MI
  2. Death caused by sudden cardiac, including unwitnessed, death
  3. Death resulting from heart failure
  4. Death caused by stroke
  5. Death caused by cardiovascular procedures
  6. Death resulting from cardiovascular hemorrhage
  7. Death resulting from other cardiovascular cause Any MI not clearly attributable to a non-target vessel will be considered as target-vessel MI.
     * Percutaneous coronary intervention (PCI) related MI is termed type 4a MI.
     * Coronary artery bypass grafting (CABG) related MI is termed type 5 MI. Revascularization is clinically driven if the target lesion diameter stenosis is > 50% by quantitative coronary angiography (QCA) and the subject has clinical or functional ischemia which cannot be explained by another native coronary or bypass graft lesion.
Bleeding | 2 year
  Bleeding BARC 2 or greater

OTHER OUTCOMES:
Composite of cardiovascular death, target vessel MI and ischemia-driven TLR (TLF) | 2 year FU
  Cardiovascular death is defined as death resulting from cardiovascular causes. Any MI not clearly attributable to a non-target vessel will be considered as target-vessel MI.
  Revascularization is clinically driven if the target lesion diameter stenosis is > 50% by quantitative coronary angiography (QCA) and the subject has clinical or functional ischemia which cannot be explained by another native coronary or bypass graft lesion.
Occurrence of cardiovascular death and target-vessel myocardial infarction (MI) | 2 year
  Cardiovascular death is defined as death resulting from cardiovascular causes. The following categories may be collected:
  1. Death caused by acute MI
  2. Death caused by sudden cardiac, including unwitnessed, death
  3. Death resulting from heart failure
  4. Death caused by stroke
  5. Death caused by cardiovascular procedures
  6. Death resulting from cardiovascular hemorrhage
  7. Death resulting from other cardiovascular cause. Any MI not clearly attributable to a non-target vessel will be considered as target-vessel MI.
     * Percutaneous coronary intervention (PCI) related MI is termed type 4a MI.
     * Coronary artery bypass grafting (CABG) related MI is termed type 5 MI.
All-cause mortality | up to 2 years from procedure
  all deaths are considered cardiovascular unless an alternate cause is unequivocally established, even among subjects with serious noncardiac comorbidities.
Stroke | up to 2 years from procedure
  according to Neuro-ARC stroke/TIA criteria
Stent thrombosis | 2 year
  defined for grade and timing according to the Academic Research Consortium2
Technical success | 2 year
  Technical success is defined as the ability to cross the occluded segment with both a wire and a balloon, and successfully open the artery; the restoration of antegrade TIMI flow 2 or 3 and a <30% residual stenosis. (As applies to chronic total occlusion - CTO - lesions)
Clinical procedural success | 2 year
  In the case of percutaneous intervention for obstructive lesions, procedural success is defined as the achievement of a final residual diameter stenosis < 30% by angiography at the end of the procedure (and without flow limiting arterial dissection and hemodynamically significant translesional pressure gradient) without any in-hospital major adverse events (death, acute onset of limb ischemia, need for urgent/emergent vascular surgery). The balloon inflation and/or stent placement may be preceded by use of adjunctive devices (e.g., percutaneous mechanical thrombectomy, directional or rotational atherectomy, laser, chronic total occlusion crossing device).
  Ideally, the assessment of the residual stenosis at the end of the procedure should be performed by an angiographic core laboratory.
Occurrence of ischemia-driven TLR | 2 year FU
  Revascularization is clinically driven if the target lesion diameter stenosis is > 50% by quantitative coronary angiography (QCA) and the subject has clinical or functional ischemia which cannot be explained by another native coronary or bypass graft lesion.
Target vessel revascularization (TVR) | up to 2 years
  TLR is a repeat percutaneous intervention of the target lesion or bypass surgery of the target vessel performed for restenosis or other complication of the target lesion.

CONTACTS AND LOCATIONS:
Overall Officials: Roxana Mehran, Study Chair — Mount Sinai Heart
Locations (90):
- Australia (3):
  - The Prince Charles Hospital, Chermside
  - St Vincent Hospital, Melbourne
  - The Wollongong Hospital, Wollongong
- Austria (2):
  - University Heart Center Graz, Graz
  - Kardinal Schwarzenberg Klinikum, Schwarzach im Pongau
- National Heart Foundation Hospital & Research Institute, Dhaka, Bangladesh
- Belgium (2):
  - Antwerp Cardiovascular Center Middelheim, Antwerp
  - UZ Leuven, Leuven
- Brazil (2):
  - Instituto Dante Pazzanese de Cardiologia, São Paulo
  - INSTITUTO DO CORAÇÃO - InCor University of São Paulo Medical School, São Paulo
- Czechia (2):
  - University Hospital Brno, Department of Medecine Cardiology, Brno
  - University Hospital Královské Vinohrady, Department of Medecine Cardiology, Prague
- France (8):
  - Clinique Axium, Aix-en-Provence
  - CHRU Brest, Brest
  - Clinique de Fontaine, Fontaine-lès-Dijon
  - Groupe Hospitalier Mutualiste de Grenoble, Grenoble
  - Hôpital La Timone, Service Cardiologie, Marseille
  - Hôpital Privé Jacques Cartier, Massy
  - CHU de Nîmes, Nîmes
  - Hôpital Cochin, Paris
- Germany (11):
  - Klinik für Kardiologie und Angiologie II, Herz-Zentrum Bad Krozingen, Bad Krozingen
  - Kerckhoff-Klinik GmbH Abteilung Kardiologie/Herzchirurgie, Bad Nauheim
  - Herzzentrum, Segeberger Kliniken GmbH, Bad Segeberg
  - Charite Berlin, Department of Cardiology, Campus Benjamin Franklin, Berlin
  - Helios Amper-Klinikum Dachau, Dept. of Cardiology & Pneumology, Dachau
  - Elisabeth Krankenhaus Essen, Essen
  - 121/ MVZ Hamburg, DEU, Hamburg
  - UKSH, Campus Kiel, Department of Cardiology, Kiel
  - Heart Center Leipzig, Leipzig
  - Universitaetsklinikum Tubingen, DEU, Tübingen
  - Schwarzwald Baar Klinikum Villingen-Schwenningen GmbH, Villingen-Schwenningen
- India (2):
  - Madras Medical Mission, Chennai
  - Krishna Institute of Medical Sciences, Secunderabad
- National University of Ireland, Galway Galway University Hospital, Galway, Ireland
- Italy (15):
  - IRCCS - Policlinico San Donato, San Donato Milanese, Milano
  - GVM - Cotignola, Cotignola, Ravenna
  - Fondazione Poliambulanza di Brescia, Brescia
  - P.O. G. Rodolico, Catania
  - 075/ Magna Graecia University, Catanzaro
  - Casa di Cura Montevergine, Mercogliano
  - Istituto Sant'Ambrogio, Milan
  - San Carlo Clinic, Milan
  - San Raffaele Hospital, Milan
  - 133/Clinica Mederranea, Napoli
  - Division of Cardiology, University of Campania "Luigi Vanvitelli", Napoli
  - 156/ Policlinico San Matteo, Pavia
  - Ospedale degli infermi, Rivoli
  - Azienda Ospedaliera San Camillo Forlanini, Roma
  - Policlinico Umberto I, "Sapienza" University of Rome Dept.of Cardiovascular, Respiratory, Nephrologic & Anesthesiologic Sciences, Roma
- Institut Jantung Negara, Kuala Lumpur, Malaysia
- Mexico (3):
  - Instituto nacional de cardiologia ignacio chavez, Mexico City
  - Grupo Intervención San Luis - Hospital de Especialidades de la Salud - San Luis Potosí City, San Luis Potosí City
  - IMSS Hospital de Especialidades UMAE 71, Torreón
- Netherlands (2):
  - Amsterdam UMC, Amsterdam
  - Maasstad Hospital, Rotterdam
- Poland (14):
  - XII Oddział Kardiologiczny PAKS w Bełchatowie, Bełchatów
  - Polsko-Amerykańskie Kliniki Serca III Oddział Kardiologii Inwazyjnej, Angiologii i Elektrokardiologii, Bielsko-Biala
  - MCSN AHoP Chrzanow, Chrzanów
  - Zgierskie Centrum Kardiologii Med-Pro Polsko-Amerykańskie Kliniki Serca, Dąbrowa Górnicza
  - American Heart of Poland, Kędzierzyn-Koźle
  - University Hospital Krakow, Krakow
  - Miedziowe Centrum Zdrowia SA, Lubin
  - Nyskie Centrum Kardiologiczne Polsko-Amerykańskich Klinik Serca w Nysie, Nysa
  - Centrum Kardiologii Inwazyjnej, Elektroterapii i Angiologii w Pińczowie, Pińczów
  - Szpital Kliniczny Przemienienia Pańskiego, Poznan
  - Oddział Kardiologii Szpitale Polskie Sztum, Sztum
  - X Department of Invasive Cardiology, Tychy American Heart of Poland SA, Tychy
  - I Oddział Kardiologii AHoP, Ustroń
  - Department of Interventional Cardiology Med-Pro American Heart of Poland, Zgierz
- Changi General Hospital, Singapore, Singapore
- Gachon University Gil Medical Center, Incheon, South Korea
- Sweden (2):
  - Örebro Univ. Hospital, Dpt. of cardiology, Örebro
  - Uppsala University hosp, Uppsala
- Switzerland (4):
  - Cardiocentro Ticino, Lugano
  - Hôpital de La Tour, Meyrin
  - Triemli Hospital, Zurich
  - University Hospital Zürich, Zurich
- Taiwan (2):
  - National Cheng Kung University Hospital, Tainan
  - Mackay Memorial Hospital, Taipei
- United Kingdom (11):
  - Belfast Health and Social Care Trust, Belfast
  - Royal blackburn hospital, Blackburn
  - The Royal Bournemouth Hospital, Bournemouth
  - Brighton & Sussex University NHS Hospitals Trust, Brighton
  - Golden Jubilee National Hospital, Clydebank
  - Craigavon Area Hospital, Craigavon
  - Ninewells Hospital, Dundee
  - King's College Hospital NHS Foundation Trust, London
  - Royal Free Hopsital, London
  - Freeman Hospital, Newcastle upon Tyne
  - Worcestershire Acute NHS Trust, Worcestershire Royal Hospital, Worcester

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] International Diabetes Federation 2015. IDF DIABETES ATLAS Seventh Edition. 2015; ISBN: 978-2-930229-81-2
- [Background] Thiele H, Zeymer U. Chapter: Cardiogenic shock in patients with acute coronary syndromes (p. 441), The ESC Textbook of Intensive and Acute Cardiovascular Care (2 ed.) [IACC]. Edited by Marco Tubaro, Pascal Vranckx, Susanna Price, and Christiaan Vrints. Updated on 22 February 2018 DOI: 10.1093/med/9780199687039.003.0049_update_003
- [Result] Kereiakes DJ, Cutlip DE, Applegate RJ, Wang J, Yaqub M, Sood P, Su X, Su G, Farhat N, Rizvi A, Simonton CA, Sudhir K, Stone GW. Outcomes in diabetic and nondiabetic patients treated with everolimus- or paclitaxel-eluting stents: results from the SPIRIT IV clinical trial (Clinical Evaluation of the XIENCE V Everolimus Eluting Coronary Stent System). J Am Coll Cardiol. 2010 Dec 14;56(25):2084-9. doi: 10.1016/j.jacc.2010.10.006. PMID 21144968
- [Result] Kufner S, Byrne RA, Dommasch M, Massberg S, Schoemig A, Kastrati A. Comparison of "limus"-eluting stents with permanent-vs biodegradable polymer in patients with diabetes mellitus with coronary artery disease. Eur Heart J 2012; 33: 558-9
- [Result] Stone GW, Kedhi E, Kereiakes DJ, Parise H, Fahy M, Serruys PW, Smits PC. Differential clinical responses to everolimus-eluting and Paclitaxel-eluting coronary stents in patients with and without diabetes mellitus. Circulation. 2011 Aug 23;124(8):893-900. doi: 10.1161/CIRCULATIONAHA.111.031070. Epub 2011 Aug 8. PMID 21824922
- [Result] Cutlip DE, Chhabra AG, Baim DS, Chauhan MS, Marulkar S, Massaro J, Bakhai A, Cohen DJ, Kuntz RE, Ho KK. Beyond restenosis: five-year clinical outcomes from second-generation coronary stent trials. Circulation. 2004 Sep 7;110(10):1226-30. doi: 10.1161/01.CIR.0000140721.27004.4B. Epub 2004 Aug 30. PMID 15337693
- [Result] Lee TT, Feinberg L, Baim DS, Holmes DR, Aroesty JM, Carrozza JP Jr, Cohen DJ, Ho KK, Cutlip DE. Effect of diabetes mellitus on five-year clinical outcomes after single-vessel coronary stenting (a pooled analysis of coronary stent clinical trials). Am J Cardiol. 2006 Sep 15;98(6):718-21. doi: 10.1016/j.amjcard.2006.03.059. Epub 2006 Jul 13. PMID 16950169
- [Result] Morgan KP, Kapur A, Beatt KJ. Anatomy of coronary disease in diabetic patients: an explanation for poorer outcomes after percutaneous coronary intervention and potential target for intervention. Heart. 2004 Jul;90(7):732-8. doi: 10.1136/hrt.2003.021014. PMID 15201238
- [Result] Hadi HA, Suwaidi JA. Endothelial dysfunction in diabetes mellitus. Vasc Health Risk Manag. 2007;3(6):853-76. PMID 18200806
- [Result] Schalkwijk CG, Stehouwer CD. Vascular complications in diabetes mellitus: the role of endothelial dysfunction. Clin Sci (Lond). 2005 Aug;109(2):143-59. doi: 10.1042/CS20050025. PMID 16033329
- [Result] Dangas GD, Claessen BE, Caixeta A, Sanidas EA, Mintz GS, Mehran R. In-stent restenosis in the drug-eluting stent era. J Am Coll Cardiol. 2010 Nov 30;56(23):1897-907. doi: 10.1016/j.jacc.2010.07.028. PMID 21109112
- [Result] Lightell DJ Jr, Woods TC. Relative resistance to Mammalian target of rapamycin inhibition in vascular smooth muscle cells of diabetic donors. Ochsner J. 2013 Spring;13(1):56-60. PMID 23532775
- [Result] Denardo SJ, Carpinone PL, Vock DM, Batich CD, Pepine CJ. Changes to polymer surface of drug-eluting stents during balloon expansion. JAMA. 2012 May 23;307(20):2148-50. doi: 10.1001/jama.2012.4111. No abstract available. PMID 22618916
- [Result] Popma JJ, Leon MB, Moses JW, Holmes DR Jr, Cox N, Fitzpatrick M, Douglas J, Lambert C, Mooney M, Yakubov S, Kuntz RE; SIRIUS Investigators. Quantitative assessment of angiographic restenosis after sirolimus-eluting stent implantation in native coronary arteries. Circulation. 2004 Dec 21;110(25):3773-80. doi: 10.1161/01.CIR.0000150331.14687.4B. Epub 2004 Dec 13. PMID 15596568
- [Result] Mulukutla SR, Vlachos HA, Marroquin OC, Selzer F, Holper EM, Abbott JD, Laskey WK, Williams DO, Smith C, Anderson WD, Lee JS, Srinivas V, Kelsey SF, Kip KE. Impact of drug-eluting stents among insulin-treated diabetic patients: a report from the National Heart, Lung, and Blood Institute Dynamic Registry. JACC Cardiovasc Interv. 2008 Apr;1(2):139-47. doi: 10.1016/j.jcin.2008.02.005. PMID 19212456
- [Result] Stenestrand U, James SK, Lindback J, Frobert O, Carlsson J, Schersten F, Nilsson T, Lagerqvist B; SCAAR/SWEDEHEART study group. Safety and efficacy of drug-eluting vs. bare metal stents in patients with diabetes mellitus: long-term follow-up in the Swedish Coronary Angiography and Angioplasty Registry (SCAAR). Eur Heart J. 2010 Jan;31(2):177-86. doi: 10.1093/eurheartj/ehp424. Epub 2009 Nov 10. PMID 19903684
- [Result] Maeng M, Jensen LO, Galloe AM, Thayssen P, Christiansen EH, Hansen KN, Helqvist S, Botker HE, Lassen JF, Thuesen L. Comparison of the sirolimus-eluting versus paclitaxel-eluting coronary stent in patients with diabetes mellitus: the diabetes and drug-eluting stent (DiabeDES) randomized angiography trial. Am J Cardiol. 2009 Feb 1;103(3):345-9. doi: 10.1016/j.amjcard.2008.09.084. Epub 2008 Nov 12. PMID 19166687
- [Result] Dibra A, Kastrati A, Mehilli J, Pache J, Schuhlen H, von Beckerath N, Ulm K, Wessely R, Dirschinger J, Schomig A; ISAR-DIABETES Study Investigators. Paclitaxel-eluting or sirolimus-eluting stents to prevent restenosis in diabetic patients. N Engl J Med. 2005 Aug 18;353(7):663-70. doi: 10.1056/NEJMoa044372. Epub 2005 Aug 16. PMID 16105990
- [Result] Stone GW, Midei M, Newman W, Sanz M, Hermiller JB, Williams J, Farhat N, Mahaffey KW, Cutlip DE, Fitzgerald PJ, Sood P, Su X, Lansky AJ; SPIRIT III Investigators. Comparison of an everolimus-eluting stent and a paclitaxel-eluting stent in patients with coronary artery disease: a randomized trial. JAMA. 2008 Apr 23;299(16):1903-13. doi: 10.1001/jama.299.16.1903. PMID 18430909
- [Result] Mahmud E, Ormiston JA, Turco MA, Popma JJ, Weissman NJ, O'Shaughnessy CD, Mann T, Hall JJ, McGarry TF, Cannon LA, Webster MW, Mandinov L, Baim DS. TAXUS Liberte attenuates the risk of restenosis in patients with medically treated diabetes mellitus: results from the TAXUS ATLAS program. JACC Cardiovasc Interv. 2009 Mar;2(3):240-52. doi: 10.1016/j.jcin.2008.12.009. PMID 19463432
- [Result] Serruys PW, Ruygrok P, Neuzner J, Piek JJ, Seth A, Schofer JJ, Richardt G, Wiemer M, Carrie D, Thuesen L, Boone E, Miquel-Herbert K, Daemen J. A randomised comparison of an everolimus-eluting coronary stent with a paclitaxel-eluting coronary stent:the SPIRIT II trial. EuroIntervention. 2006 Nov;2(3):286-94. PMID 19755303
- [Result] Grube E, Chevalier B, Guagliumi G, Smits PC, Stuteville M, Dorange C, Papeleu P, Kaul U, Dzavik V. The SPIRIT V diabetic study: a randomized clinical evaluation of the XIENCE V everolimus-eluting stent vs the TAXUS Liberte paclitaxel-eluting stent in diabetic patients with de novo coronary artery lesions. Am Heart J. 2012 May;163(5):867-875.e1. doi: 10.1016/j.ahj.2012.02.006. Epub 2012 Apr 11. PMID 22607866
- [Result] Garcia-Garcia HM, McFadden EP, Farb A, Mehran R, Stone GW, Spertus J, Onuma Y, Morel MA, van Es GA, Zuckerman B, Fearon WF, Taggart D, Kappetein AP, Krucoff MW, Vranckx P, Windecker S, Cutlip D, Serruys PW; Academic Research Consortium. Standardized End Point Definitions for Coronary Intervention Trials: The Academic Research Consortium-2 Consensus Document. Eur Heart J. 2018 Jun 14;39(23):2192-2207. doi: 10.1093/eurheartj/ehy223. PMID 29897428
- [Result] Thygesen K, Alpert JS, Jaffe AS, Chaitman BR, Bax JJ, Morrow DA, White HD; Executive Group on behalf of the Joint European Society of Cardiology (ESC)/American College of Cardiology (ACC)/American Heart Association (AHA)/World Heart Federation (WHF) Task Force for the Universal Definition of Myocardial Infarction. Fourth Universal Definition of Myocardial Infarction (2018). J Am Coll Cardiol. 2018 Oct 30;72(18):2231-2264. doi: 10.1016/j.jacc.2018.08.1038. Epub 2018 Aug 25. No abstract available. PMID 30153967
- [Result] Lansky AJ, Messe SR, Brickman AM, Dwyer M, van der Worp HB, Lazar RM, Pietras CG, Abrams KJ, McFadden E, Petersen NH, Browndyke J, Prendergast B, Ng VG, Cutlip DE, Kapadia S, Krucoff MW, Linke A, Moy CS, Schofer J, van Es GA, Virmani R, Popma J, Parides MK, Kodali S, Bilello M, Zivadinov R, Akar J, Furie KL, Gress D, Voros S, Moses J, Greer D, Forrest JK, Holmes D, Kappetein AP, Mack M, Baumbach A. Proposed Standardized Neurological Endpoints for Cardiovascular Clinical Trials: An Academic Research Consortium Initiative. J Am Coll Cardiol. 2017 Feb 14;69(6):679-691. doi: 10.1016/j.jacc.2016.11.045. PMID 28183511
- [Result] Mehran R, Rao SV, Bhatt DL, Gibson CM, Caixeta A, Eikelboom J, Kaul S, Wiviott SD, Menon V, Nikolsky E, Serebruany V, Valgimigli M, Vranckx P, Taggart D, Sabik JF, Cutlip DE, Krucoff MW, Ohman EM, Steg PG, White H. Standardized bleeding definitions for cardiovascular clinical trials: a consensus report from the Bleeding Academic Research Consortium. Circulation. 2011 Jun 14;123(23):2736-47. doi: 10.1161/CIRCULATIONAHA.110.009449. No abstract available. PMID 21670242
- [Derived] Abizaid A, Mehran R, Oliva A, Chamie D, Staico R, Malik F, Vink M, Kurniadi A, Cao D, Capranzano P, Faurie B, Garot P, Hildick-Smith D, Ielasi A, Loffelhardt N, Kedev S, Mylotte D, Milewski K, Paradies V, Schmitz T, Teeuwen K, Testa L, Toelg R, Vochelet F, Vogel B, Wykrzykowska J, Sartori S, Colombo A, Saito S, Morice MC; ABILITY Diabetes Global investigators. Abluminus DES+ sirolimus-eluting stent versus everolimus-eluting stent in patients with diabetes and coronary artery disease (ABILITY Diabetes Global): results from a multicentre, randomised controlled trial. Lancet. 2026 Jan 8:S0140-6736(25)02157-9. doi: 10.1016/S0140-6736(25)02157-9. Online ahead of print. PMID 41520674